CLINICAL TRIAL: NCT05388240
Title: Mobile App for Shoulder Rehabilitation Following Breast Reconstruction: A Pilot Study
Brief Title: Shoulder Rehabilitation Using a Mobile App Following Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Principal Investigator, Soo Kim, Associate Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bio2738
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Shoulder Dysfunction; Breast Reconstruction
Keywords: Mobile App
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Randomized control trial; pilot study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Active Comparator): The Education Group will be provided with standard education by the physiotherapist at the hospital prior to surgery and will be advised to continue with their normal activities of daily living (ADL). They will have access to the "standard education and resources" tabs on the mobile app. Shoulder specific exercises tab on the app will be available to them upon their completion of the study (eight weeks post-intervention).
  Interventions: Other: Education via a Mobile App
- Education plus Exercise Group (Experimental): The Exercise plus Education Group will be provided with standard education by the physiotherapist at the hospital prior to surgery. Participants in this group will have access to the "education and resources" tabs on the app.
  Interventions: Other: Education and Exercise via a Mobile App

INTERVENTIONS:
Other: Education via a Mobile App — This group will have access to "Education and Resources" tab that includes customary information given at a pre-op appointment plus some additional related education and resources.
  Arms: Education Group
Other: Education and Exercise via a Mobile App — This group will have access to "Education and Resources" tab that includes customary information given at a pre-op appointment plus some additional related education and resources. The app will also be used to help guide participants through an eight-week shoulder exercise program, together with physical therapy remote support.
  Arms: Education plus Exercise Group

SUMMARY:
Breast cancer is the most common cancer for Canadian women. Of the women who will have a mastectomy each year in Canada, one in five will elect to have breast reconstruction. However, the significant benefits for body-image, self-esteem, sexuality, and quality of life are tempered by post-treatment shoulder dysfunction for many. As a means to decrease shoulder morbidities in breast cancer survivors (BCS), this study will introduce a mobile application (app)-based shoulder rehabilitation program as an option to improve functional outcomes of the shoulder, for those who have had breast reconstruction.

DETAILED DESCRIPTION:
The percentage of Canadian women surviving at least 5 years beyond initial diagnosis is currently approaching 90% and many of these women are choosing to have breast reconstruction following mastectomy. Potential sequelae from both mastectomy and all types of breast reconstruction surgeries can result in various functional limitations. The most common adverse effect from breast cancer surgery is shoulder morbidity, having both short and long-term consequences for survivors, and evidence suggests women who undergo breast reconstruction are at even higher risk of developing shoulder problems. Shoulder/arm pain, reductions in strength, and limitations in range of motion (ROM) are some of the common physical issues plaguing BCS, often for years after the initial treatment. Fibrosis of the direct area of the target tissue is a common finding post radiation therapy, specifically of the anterior chest/ pectoralis and axilla regions in BCS and most noticeable starting six months post-surgically.

The researchers' interest in the feasibility of a shoulder rehabilitation mobile app for post-surgical BCS is to improve access to rehabilitation (including education, exercises, and remote support with a physical therapist, PT) for these women, allowing for better functional outcomes which could translate into decreased reliance on medical care, improved quality of life (QoL), and ability to participate in life roles.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years of age
* scheduled for immediate or delayed breast reconstruction (implant type only)
* 6 weeks or less from time of surgery
* must have mobile phone capable of app download
* need desk top or laptop computer for Zoom meetings
* medically stable
* able to be informed and consent in English

Exclusion Criteria:

* ongoing or current health-related issues that would interfere with the ability to complete the program (i.e. metastatic cancer, severe cardiovascular disease)
* lack of access to a mobile phone and laptop or desk top computer for Zoom meetings
* inability to comprehend the English language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Shoulder Range of Motion (ROM) | At start of the study, at 4 weeks into the study and again at the end of the study (8 weeks into the study).
  ROM measurements of both shoulders (flexion, extension, abduction, internal and external rotation) will be taken post-operatively, via the downloaded app on each participant's phone, and by visual examination of the research assistant (registered, licensed PT) during the virtual assessment via Zoom. These ROM measures, taken at the beginning of the intervention (week one), mid-intervention (week four), and end of intervention (week eight) will be used as a guide for exercise progression throughout the intervention. The measurements will also be used in our data analysis to understand changes in shoulder ROM from the beginning of the intervention to the end of intervention.

SECONDARY OUTCOMES:
Quick Disability of Arm, Shoulder and Hand (Quick DASH) | At start of the study, at 4 weeks into the study and again at the end of the study (8 weeks into the study).
  The Quick DASH is an 11-item questionnaire measuring perceived upper extremity functional ability as well as symptoms on a 5-point scale from 1 (no difficulty) to 5 (unable) (Budtz, 2018). The Quick DASH is quick and easy to administer and to score, and has been used to measure shoulder function in the BCS population in previous studies (Chan et al., 2020; Duymaz et al., 2019; Lang et al., 2020). Data from this questionnaire will be used to better understand changes in upper extremity functional ability and symptoms from the start to end of intervention.
Visual Analogue Scale (VAS) | At start of the study, at 4 weeks into the study and again at the end of the study (8 weeks into the study).
  The VAS is a tool measuring intensity of symptoms from 0 (no pain) to 10 (worst pain). Each participant will be asked to rate their current shoulder pain on the continuum of this tool and this rating will be used to understand the level of shoulder pain of each participant on the day of assessment. Pain levels from start of intervention, to mid-intervention (at four weeks), to end of intervention (at eight weeks), will be analyzed using continuous ordinal regression or normal-distribution methods (t-test, linear regression) depending on the data collected, and to best understand significance of changes in pain levels from beginning to end of the intervention (Heller et al., 2016). Because of its simplicity and ease of use, it can be administered broadly across a wide variety of populations and can be presented in multiple ways, targeting certain populations of interest (Wewers et al., 1990).
Fatigue Assessment Scale (FAS) | At start of the study, at 4 weeks into the study and again at the end of the study (8 weeks into the study).
  The FAS is a 10-item questionnaire, that measures fatigue symptoms on a 5-point scale from "Never" (1) to "Always" (5). Although the development and use of most fatigue scales, including the FAS, have been disease specific, most often they have been developed to assess fatigue in people with cancer (Hjollund, 2007). The FAS will be analyzed similarly to the VAS to best understand significance of changes in fatigue levels from beginning to end of intervention.
Short Form 36 (SF-36) | At start of the study, at 4 weeks into the study and again at the end of the study (8 weeks into the study).
  The SF-36 is a 36-question survey aimed at measuring quality of life (QoL). This tool has been well researched and highly used in all populations, including healthy and disease specific populations (Ware et al., 1992), as well as in research (Ware et al., 1992; Lins et al., 2016). Reliability of the SF-36 is good for several diagnoses, including adult survivors of childhood cancer (Reulen, 2006). As the SF-36 measures both physical and mental health, research suggests its use in combination with other outcome measures when assessing overall QoL (Lins et al., 2016), hence the inclusion of other outcome measures as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Kim, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canadian Cancer Statistics 2019. Toronto, ON. (2019). Retrieved November 30, 2020 from http://www.cancer.ca/~/media/cancer.ca/CW/cancer information/cancer 101/Canadian cancer statistics/Canadian-Cancer-Statistics 2019-EN.pdf?la=en.
- [Background] Ditsch N, Bauerfeind I, Vodermaier A, Tripp C, Lohrs B, Toth B, Himsl I, Graeser M, Harbeck N, Lenhard M. A retrospective investigation of women's experience with breast reconstruction after mastectomy. Arch Gynecol Obstet. 2013 Mar;287(3):555-61. doi: 10.1007/s00404-012-2590-1. Epub 2012 Oct 23. PMID 23090185
- [Background] Zhong T, Hu J, Bagher S, Vo A, O'Neill AC, Butler K, Novak CB, Hofer SOP, Metcalfe KA. A Comparison of Psychological Response, Body Image, Sexuality, and Quality of Life between Immediate and Delayed Autologous Tissue Breast Reconstruction: A Prospective Long-Term Outcome Study. Plast Reconstr Surg. 2016 Oct;138(4):772-780. doi: 10.1097/PRS.0000000000002536. PMID 27673514
- [Background] Nesvold IL, Fossa SD, Holm I, Naume B, Dahl AA. Arm/shoulder problems in breast cancer survivors are associated with reduced health and poorer physical quality of life. Acta Oncol. 2010 Apr;49(3):347-53. doi: 10.3109/02841860903302905. PMID 19842790
- [Background] Blackburn NE, Mc Veigh JG, Mc Caughan EM, Kennedy RD, McIntosh SA, Wilson IM. The musculoskeletal consequences of latissmus dorsi breast reconstruction in women following mastectomy for breast cancer. PLoS One. 2018 Aug 28;13(8):e0202859. doi: 10.1371/journal.pone.0202859. eCollection 2018. PMID 30153282
- [Background] Blackburn NE, Mc Veigh JG, Mc Caughan E, Wilson IM. The musculoskeletal consequences of breast reconstruction using the latissimus dorsi muscle for women following mastectomy for breast cancer: A critical review. Eur J Cancer Care (Engl). 2018 Mar;27(2):e12664. doi: 10.1111/ecc.12664. Epub 2017 Feb 10. PMID 28185324
- [Background] Verbelen H, Tjalma W, Meirte J, Gebruers N. Long-term morbidity after a negative sentinel node in breast cancer patients. Eur J Cancer Care (Engl). 2019 Sep;28(5):e13077. doi: 10.1111/ecc.13077. Epub 2019 May 3. PMID 31050088
- [Background] Riekki R, Harvima IT, Jukkola A, Risteli J, Oikarinen A. The production of collagen and the activity of mast-cell chymase increase in human skin after irradiation therapy. Exp Dermatol. 2004 Jun;13(6):364-71. doi: 10.1111/j.0906-6705.2004.00164.x. PMID 15186323
- [Background] Karki A, Simonen R, Malkia E, Selfe J. Impairments, activity limitations and participation restrictions 6 and 12 months after breast cancer operation. J Rehabil Med. 2005 May;37(3):180-8. doi: 10.1080/16501970410024181. PMID 16040476
- [Background] Budtz CR, Andersen JH, de Vos Andersen NB, Christiansen DH. Responsiveness and minimal important change for the quick-DASH in patients with shoulder disorders. Health Qual Life Outcomes. 2018 Dec 10;16(1):226. doi: 10.1186/s12955-018-1052-2. PMID 30526622
- [Background] Chan KS, Zeng D, Leung JHT, Ooi BSY, Kong KT, Yeo YH, Goo JTT, Chia CLK. Measuring upper limb function and patient reported outcomes after major breast cancer surgery: a pilot study in an Asian cohort. BMC Surg. 2020 May 19;20(1):108. doi: 10.1186/s12893-020-00773-0. PMID 32430021
- [Background] Duymaz T, Iyigun ZE, Ilgun AS, Ordu C, Ucuncu M, Alco G, Ozturk A, Elbuken F, Aktepe F, Ozmen V. The Effect of Mini-Latissimus Dorsi Flap (MLDF) Reconstruction on Shoulder Function in Breast Cancer Patients. Eur J Breast Health. 2019 Jul 1;15(3):158-162. doi: 10.5152/ejbh.2019.4727. eCollection 2019 Jul. PMID 31312791
- [Background] Lang, A. (2020). Towards Improving Clinical Evaluation of the Shoulder: Defining Upper Limb Biomechanics of Breast Cancer Survivors During Functional Evaluation Tasks (Doctoral Dissertation). University of Saskatchewan.
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536
- [Background] Hjollund NH, Andersen JH, Bech P. Assessment of fatigue in chronic disease: a bibliographic study of fatigue measurement scales. Health Qual Life Outcomes. 2007 Feb 27;5:12. doi: 10.1186/1477-7525-5-12. PMID 17326844
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230
- [Background] Reulen RC, Zeegers MP, Jenkinson C, Lancashire ER, Winter DL, Jenney ME, Hawkins MM. The use of the SF-36 questionnaire in adult survivors of childhood cancer: evaluation of data quality, score reliability, and scaling assumptions. Health Qual Life Outcomes. 2006 Oct 5;4:77. doi: 10.1186/1477-7525-4-77. PMID 17022814
- [Background] Lee, S. (2021). Breast cancer statistics. Canadian Cancer Society. Retrieved March 9, 2022, from https://cancer.ca/en/cancer-information/cancer-types/breast/statistics
- [Background] Plastic surgery statistics. American Society of Plastic Surgeons. (2020). Retrieved March 9, 2022, from https://www.plasticsurgery.org/news/plastic-surgery-statistics
- [Background] Ware, J. E. (1993, January). SF-36 Health Survey: Manual & Interpretation Guide. ResearchGate. https://www.researchgate.net/publication/313050850_SF-36_Health_Survey_Manual_Interpretation_Guide